CLINICAL TRIAL: NCT01463917
Title: Use of Hypertonic Versus Isotonic Solutions in Off Pump Coronary Artery Bypass Graft Surgery Targeting the Left Marginal Branch
Brief Title: Hypertonic Solution in Off Pump Coronary Artery Bypass Graft Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Pitangueiras (Other)
Responsible Party: Principal Investigator, Roberto Rocha e Silva, Chief, Adult Heart Surgery, MD PHD in Cardiovascular Surgery, Hospital Pitangueiras
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: hypertonic off pump CABS
Record Dates: First submitted 2011-10-19; First posted 2011-11-02 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-10

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Bypass; Off-Pump; Saline Solution; Hypertonic
MeSH Terms: conditions — Coronary Artery Disease | interventions — Hypertonic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypertonic (Active Comparator): Use of Hypertonic solution during left marginal branch CABG surgery.
  Interventions: Drug: Hypertonic solution
- Isotonic (Placebo Comparator): Use of Isotonic solution during left marginal branch CABG surgery.
  Interventions: Drug: Isotonic

INTERVENTIONS:
Drug: Hypertonic solution — Use of Hypertonic solution 4 ml/Kg during left marginal branch CABG surgery.
  Arms: Hypertonic
Drug: Isotonic — Use of Isotonic solution 4 ml/Kg during left marginal branch CABG surgery.
  Arms: Isotonic

SUMMARY:
This is a comparison between Hypertonic versus isotonic solution in a double blind randomized trial for off pump Coronary Artery Bypass Graft (CABG) surgery targeting the left marginal branch.

Hypertonic solution should provide better tolerance for heart mobilization with less volume expansion and less drugs.

ELIGIBILITY:
Inclusion Criteria:

* Off pump CABG targeting the left marginal branch

Exclusion Criteria:

* On pump surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-03 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Use of vasoactive drugs in left marginal branch off pump CABG surgery | time related to left branch coronary anastomosis for drug need.
  Comparison between hypertonic and isotonic solutions for need of vasoactive drugs with heart mobilization during left marginal branch off pump CABG surgery. Data will be collected respectively at 1, 5 and 10 minutes after beggining the left branch coronary anastomosis. Data will be type of drug need and dosage until the end os the anastomosis.

SECONDARY OUTCOMES:
Fluid balance | Operative period and first operative day
  Comparison of fluid balance in the operative period between hypertonic and isotonic solutions. Data will be collected at the end of surgery and by next mornning.

CONTACTS AND LOCATIONS:
Overall Officials: ROBERTO R Silva, MD PHD, Principal Investigator — Hospital Pitangueiras
Locations (1):
- Hospital Pitangueiras, Jundiaí, São Paulo, Brazil

REFERENCES:
- [Background] Velasco IT, Pontieri V, Rocha e Silva M Jr, Lopes OU. Hyperosmotic NaCl and severe hemorrhagic shock. Am J Physiol. 1980 Nov;239(5):H664-73. doi: 10.1152/ajpheart.1980.239.5.H664. PMID 6776826
- [Background] Rocha e Silva M, Braga GA, Prist R, Velasco IT, Granca ES. Isochloremic hypertonic solutions for severe hemorrhage. J Trauma. 1993 Aug;35(2):200-5. doi: 10.1097/00005373-199308000-00005. PMID 7689115
- [Background] Wade CE, Kramer GC, Grady JJ, Fabian TC, Younes RN. Efficacy of hypertonic 7.5% saline and 6% dextran-70 in treating trauma: a meta-analysis of controlled clinical studies. Surgery. 1997 Sep;122(3):609-16. doi: 10.1016/s0039-6060(97)90135-5. PMID 9308620
- [Background] Mazzoni MC, Borgstrom P, Intaglietta M, Arfors KE. Capillary narrowing in hemorrhagic shock is rectified by hyperosmotic saline-dextran reinfusion. Circ Shock. 1990 Aug;31(4):407-18. PMID 1697790
- [Background] Ramires JA, Serrano Junior CV, Cesar LA, Velasco IT, Rocha e Silva Junior M, Pileggi F. Acute hemodynamic effects of hypertonic (7.5%) saline infusion in patients with cardiogenic shock due to right ventricular infarction. Circ Shock. 1992 Jul;37(3):220-5. PMID 1423912
- [Background] Auler JO Jr, Pereira MH, Gomide-Amaral RV, Stolf NG, Jatene AD, Rocha e Silva M. Hemodynamic effects of hypertonic sodium chloride during surgical treatment of aortic aneurysms. Surgery. 1987 May;101(5):594-601. PMID 3576451
- [Background] DeFoe GR, Ross CS, Olmstead EM, Surgenor SD, Fillinger MP, Groom RC, Forest RJ, Pieroni JW, Warren CS, Bogosian ME, Krumholz CF, Clark C, Clough RA, Weldner PW, Lahey SJ, Leavitt BJ, Marrin CA, Charlesworth DC, Marshall P, O'Connor GT. Lowest hematocrit on bypass and adverse outcomes associated with coronary artery bypass grafting. Northern New England Cardiovascular Disease Study Group. Ann Thorac Surg. 2001 Mar;71(3):769-76. doi: 10.1016/s0003-4975(00)02393-6. PMID 11269449
- [Background] Boldt J, Zickmann B, Ballesteros M, Herold C, Dapper F, Hempelmann G. Cardiorespiratory responses to hypertonic saline solution in cardiac operations. Ann Thorac Surg. 1991 Apr;51(4):610-5. doi: 10.1016/0003-4975(91)90320-p. PMID 2012420
- [Background] Boldt J, Zickmann B, Herold C, Ballesteros M, Dapper F, Hempelmann G. Influence of hypertonic volume replacement on the microcirculation in cardiac surgery. Br J Anaesth. 1991 Nov;67(5):595-602. doi: 10.1093/bja/67.5.595. PMID 1721516 (Retraction: PMID 32861403 Br J Anaesth. 2020 Sep;125(3):412-413)
- [Background] Oliveira SA, Bueno RM, Souza JM, Senra DF, Rocha-e-Silva M. Effects of hypertonic saline dextran on the postoperative evolution of Jehovah's Witness patients submitted to cardiac surgery with cardiopulmonary bypass. Shock. 1995 Jun;3(6):391-4. PMID 7544684
- [Background] Sirieix D, Hongnat JM, Delayance S, D'Attellis N, Vicaut E, Berrebi A, Paris M, Fabiani JN, Carpentier A, Baron JF. Comparison of the acute hemodynamic effects of hypertonic or colloid infusions immediately after mitral valve repair. Crit Care Med. 1999 Oct;27(10):2159-65. doi: 10.1097/00003246-199910000-00014. PMID 10548199
- [Background] Tollofsrud S, Noddeland H. Hypertonic saline and dextran after coronary artery surgery mobilises fluid excess and improves cardiorespiratory functions. Acta Anaesthesiol Scand. 1998 Feb;42(2):154-61. doi: 10.1111/j.1399-6576.1998.tb05101.x. PMID 9509195
- [Background] Rocha-E-Silva R, Caneo LF, Lourenco Filho DD, Jatene MB, Barbero-Marcial M, Oliveira SA, Rocha-E-Silva M. First use of hypertonic saline dextran in children: a study in safety and effectiveness for atrial septal defect surgery. Shock. 2003 Nov;20(5):427-30. doi: 10.1097/01.SHK.0000094037.09886.d2. PMID 14560106
- [Background] Kvalheim VL, Farstad M, Steien E, Mongstad A, Borge BA, Kvitting PM, Husby P. Infusion of hypertonic saline/starch during cardiopulmonary bypass reduces fluid overload and may impact cardiac function. Acta Anaesthesiol Scand. 2010 Apr;54(4):485-93. doi: 10.1111/j.1399-6576.2009.02156.x. Epub 2009 Oct 29. PMID 19878097
- [Background] Mustafa I, Leverve XM. Metabolic and hemodynamic effects of hypertonic solutions: sodium-lactate versus sodium chloride infusion in postoperative patients. Shock. 2002 Oct;18(4):306-10. doi: 10.1097/00024382-200210000-00003. PMID 12392272
- [Background] Chang WI, Kim KB, Kim JH, Ham BM, Kim YL. Hemodynamic changes during posterior vessel off-pump coronary artery bypass: comparison between deep pericardial sutures and vacuum-assisted apical suction device. Ann Thorac Surg. 2004 Dec;78(6):2057-62. doi: 10.1016/j.athoracsur.2004.05.059. PMID 15561035
- [Background] Ozay B, Sargin M, Abay G, Ketenci B, Kut S, Enc Y, Orhan G, Teskin O, Demirtas M. The severity of positional mitral regurgitation during off-pump coronary artery bypass grafting. Heart Surg Forum. 2008;11(3):E145-51. doi: 10.1532/HSF98.20071191. PMID 18583284
- [Background] Mishra M, Malhotra R, Mishra A, Meharwal ZS, Trehan N. Hemodynamic changes during displacement of the beating heart using epicardial stabilization for off-pump coronary artery bypass graft surgery. J Cardiothorac Vasc Anesth. 2002 Dec;16(6):685-90. doi: 10.1053/jcan.2002.128418. PMID 12486647
- [Background] Rocha-e-Silva M, Negraes GA, Soares AM, Pontieri V, Loppnow L. Hypertonic resuscitation from severe hemorrhagic shock: patterns of regional circulation. Circ Shock. 1986;19(2):165-75. PMID 3719918